CLINICAL TRIAL: NCT00483405
Title: Phase II Study of Oxaliplatin, Capecitabine, and Cetuximab in Advanced Hepatocellular Carcinoma
Brief Title: Oxaliplatin, Capecitabine, and Cetuximab in Treating Patients With Advanced Liver Cancer
Acronym: NRR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Sanofi (Industry); Roche Pharma AG (Industry); Bristol-Myers Squibb (Industry); National Center for Research Resources (NCRR) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0421; KL2RR025746 (NIH); 5K23CA118431-02 (NIH)
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Liver Cancer
Keywords: advanced adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Cetuximab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Trial (Other): Single Arm Trial
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Biological: cetuximab — 250 mg/m2, intravenously, once per week
  Other Names: Erbitux
Drug: capecitabine — 850 mg/m2, orally, twice daily (dose rounded to accommodate 150 mg and 500 mg tablet sizes. Capecitabine given on days 1-14 of 21 day cycle.
  Other Names: Xeloda
Drug: oxaliplatin — 130 mg/m2, intravenously on Day 1 of each 21 day cycle
  Other Names: Eloxatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving chemotherapy together with a monoclonal antibody may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving oxaliplatin and capecitabine together with cetuximab works in treating patients with advanced liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with advanced hepatocellular carcinoma and hepatic dysfunction treated with oxaliplatin, capecitabine, and cetuximab.

Secondary

* Determine the safety of this regimen in these patients.
* Determine the overall survival of patients treated with this regimen.
* Determine the time to tumor progression in patients treated with this regimen.

OUTLINE: This is an open label, nonrandomized study.

Patients receive oral capecitabine twice daily on days 1-14, cetuximab IV over 60-120 minutes on days 1, 8, and 15, and oxaliplatin IV over 120 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 3-4 weeks and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Histologically confirmed hepatocellular carcinoma
  * Alpha-fetoprotein (AFP) > 400 ng/mL with compatible mass by CT scan or MRI
* Metastatic disease OR not a candidate for surgical resection or immediate liver transplantation
* At least 1 site of measurable disease OR evaluable disease (AFP 2 times upper limit of normal (ULN))
* No evidence of central nervous system (CNS) metastases (unless CNS metastases stable for > 3 months)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 3 times ULN
* International normalized ratio (INR) ≤ 1.5
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times ULN
* Creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to capecitabine, cetuximab, or oxaliplatin or to other murine products
* No comorbid condition which is deemed by the investigator to have a life expectancy of < 6 months
* No New York Heart Association class III-IV coronary artery disease and/or heart failure
* No variceal bleeding within the past 60 days
* No other cancer within the past 5 years except cervical intraepithelial neoplasia, nonmelanoma skin cancer, ductal carcinoma in situ, chronic lymphocytic leukemia, or treated localized prostate cancer with a normal prostate specific antigen level
* No active drug or alcohol abuse
* No prior allergic reaction to a therapeutic antibody
* No serious, uncontrolled infection
* No history of uncontrolled seizures, CNS disorders, or psychiatric disability that, in the opinion of the investigator, would preclude study participation or compliance
* No other serious uncontrolled medical condition that, in the opinion of the investigator, would preclude study participation
* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome
* No known existing uncontrolled coagulopathy

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior participation in an investigational drug trial
* At least 4 weeks since prior major surgery and recovered
* At least 4 weeks since prior embolization, resection, or ablation
* No prior epidermal growth factor receptor (EGFR)-targeting therapy
* No prior systemic chemotherapy or hepatic artery infusion of chemotherapy
* No concurrent phenytoin
* No concurrent therapeutic warfarin

  * Low-dose non-therapeutic warfarin to maintain patency of venous access devices allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-10; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Michael A. Morse, MD, Principal Investigator — Duke University
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sanoff HK, Bernard S, Goldberg RM, Morse MA, Garcia R, Woods L, Moore DT, O'Neil BH. Phase II Study of Capecitabine, Oxaliplatin, and Cetuximab for Advanced Hepatocellular Carcinoma. Gastrointest Cancer Res. 2011 May;4(3):78-83. PMID 22043322
- See also: University of North Carolina Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 33 enrolled; 2 patients withdrew or refused prior to the beginning of protocol therapy, 2 patients were found to be ineligible, and 1 patient was withdrawn when diagnosis changed to sarcoma.
Period: Overall Study
Arm/Group | Single Arm Trial
Started | 28
Completed | 0
Not Completed | 28
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 14
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Other complicating disease | 1

BASELINE CHARACTERISTICS:
Population: 29 patients received any protocol directed therapy, but only 28 patients were included in any efficacy analysis because one patient was found to have a sarcoma and was withdrawn from the study.
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 59 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
The Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale from 0-5 to describe a patient's level of functioning in terms of self care ability and activity level.
  0. Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all self care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited self care; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self care; totally confined to bed or chair
  5. Dead
  Participants
    0 | 14
    1 | 12
    2 | 1
Childs-Pugh Classification [Count of Participants; unit: Participants] — Child-Pugh scores five clinical features and is used to assess the prognosis of chronic liver disease and cirrhosis. The lower the points total, the better prognosis. Population: Childs-Pugh was available only for the 24 evaluable patients.
  Participants
    Class A (5-6 points): number analyzed (Participants) | 24
    Class A (5-6 points) | 18
    Class B (7-9 points): number analyzed (Participants) | 24
    Class B (7-9 points) | 6
    Class C (10-15 points) | 0
Prior Therapy [Count of Participants; unit: Participants]
  Yes | 13
  None | 15

OUTCOME MEASURES:

1. Primary Outcome: Disease Response Rate
Description: Radiographic response will be measured every six weeks while subject is on treatment. Response will be measured using RECIST criteria.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 42 days (2 cycles)
Population: Four patients received some protocol treatment but withdrew before completing one cycle without assessment of response.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 24
percentage of participants with response | 12.5 [3 to 32]

2. Secondary Outcome: Number of Subjects Experiencing Adverse Events
Description: Adverse events will be assessed using CTCAE criteria.
Time Frame: every 3 weeks of treatment with an average of 15 weeks on treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 29
Participants | 29

3. Secondary Outcome: Overall Survival
Description: Overall survival will be calculated from time of enrollment to death or last contact date.
Time Frame: Median 23 month follow-up
Population: Four patients received some protocol treatment but withdrew before completing one cycle without assessment of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 24
months | 4.4 [2.4 to 7.3]

4. Secondary Outcome: Time to Progression
Description: Time to progression will be calculated from the time of enrollment until confirmed disease progression. Defined by RECIST (Response Evaluation Criteria in Solid Tumors), Progressive Disease (PD) - at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Median 23 month follow-up
Population: Four patients received some protocol treatment but withdrew before completing one cycle without assessment of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 24
months | 4.5 [3.2 to 6.4]

ADVERSE EVENTS:
Time Frame: Toxicity was assessed the second week of cycle 1 then at the commencement of each subsequent cycle.
Arm/Group | Single Arm Trial
All-Cause Mortality (participants affected / at risk) | 27/29
Serious Adverse Events (participants affected / at risk) | 17/29
Other Adverse Events (participants affected / at risk) | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=29)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2
Bilirubin (hyperbilirubinemia) (Investigations) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Conduction abnormality/atrioventricular heart block - AV Block-Third degree (Complete AV block) (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Creatinine (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Edema: limb (General disorders) | 2
Edema: viscera (General disorders) | 1
Encephalopathy (Nervous system disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 1
Hemorrhage, GI - Esophagus (Gastrointestinal disorders) | 1
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1
Hemorrhage, GI - Upper GI NOS (Gastrointestinal disorders) | 1
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 4
Infection with normal ANC or Grade 1 or 2 neutrophils - Salivary gland (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1
Leukocytes (total WBC) (Investigations) | 1
Lipase (Investigations) | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4
Renal failure (Renal and urinary disorders) | 3
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=29)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 21
Alkaline phosphatase (Investigations) | 18
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 15
Anorexia (Metabolism and nutrition disorders) | 11
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 18
Bilirubin (hyperbilirubinemia) (Investigations) | 14
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 19
Constipation (Gastrointestinal disorders) | 7
Creatinine (Investigations) | 9
Diarrhea (Gastrointestinal disorders) | 16
Fatigue (asthenia, lethargy, malaise) (General disorders) | 20
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10
Hemoglobin (Blood and lymphatic system disorders) | 15
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 6
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 14
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 24
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 18
Neuropathy: sensory (Nervous system disorders) | 20
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8
Pain - Abdomen NOS (Gastrointestinal disorders) | 9
Platelets (Blood and lymphatic system disorders) | 15
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 10
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 16
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 6
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 11
Vomiting (Gastrointestinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes